CLINICAL TRIAL: NCT00737698
Title: Is the Anaerobic Quadriceps Muscle Phenotype in Chronic Obstructive Pulmonary Disease Mediated by Reduced Muscle Concentrations of Peroxisome Proliferator-Activated Receptors Alpha and Delta?
Brief Title: Comparison of Repetitive Magnetic Stimulation and Exercise on Quadriceps Function in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); Maastricht University (Other); Magstim Company, Whitland, Wales (Unknown)
Responsible Party: Principal Investigator, Amanda Sathyapala, Wellcome Trust Clinical Research Fellow, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: rMS v exercise in COPD
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exercise; repetitive magnetic stimulation; quadriceps strength
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Experimental): Exercise
  Interventions: Other: Exercise
- Repetitive magnetic stimulation (Experimental): Repetitive magnetic stimulation of femoral nerve
  Interventions: Other: Repetitive magnetic stimulation
- Control (No Intervention): No active treatment

INTERVENTIONS:
Other: Exercise — Physiotherapist-supervised exercise course (endurance and resistance exercises) for 2 hours twice a week for 8 weeks
  Arms: Exercise
Other: Repetitive magnetic stimulation — Repetitive magnetic stimulation of the intramuscular branches of the femoral nerve for 3 hours twice a week for 8 weeks
  Arms: Repetitive magnetic stimulation

SUMMARY:
Background Chronic Obstructive Pulmonary Disease (COPD) patients develop leg weakness and a reduced walking capacity, due to reduced leg muscle oxygen-utilising capacity (OUC). Animal experiments indicate that low muscle levels of Peroxisome Proliferator-Activated Receptors (PPAR) cause the reduced muscle OUC.

Aims

In COPD patients, investigate whether:

1. reduced muscle PPAR levels cause reduced leg muscle OUC, by investigating a correlation between these in muscle samples (Study 1).
2. training increases muscle PPAR levels in proportion to increases in OUC, as should occur if PPARs control OUC (Study 2).
3. muscle PPAR levels and walking capacity correlate (Study 1 and 2).

3. the new technique of repetitive stimulation of the nerve to the leg with a magnet (rMS) improves muscle OUC (Study 2).

Study 1 Leg weakness and walking ability are assessed in 75 patients, then a leg muscle sample is taken to measure PPARs and OUC.

Study 2 60 Study 1 patients have either cardiovascular training, rMS, or no training, for 8 weeks, then are re-studied as in Study 1.

Importance If reduced PPAR levels correspond with leg weakness, medicines can be developed to target these receptors and treat weakness. If rMS is effective, it can be offered to patients.

DETAILED DESCRIPTION:
There has been considerable interest in finding methods of improving quadriceps function in COPD, since quadriceps dysfunction is associated with reduced exercise capacity5 and survival in patients16, independently of lung function. Pulmonary rehabilitation (PR) courses comprising exercise and education can increase oxidative enzymes, strength and endurance of the quadriceps in patients with COPD17 and improve walking capacity even over a period of 8 weeks12, 18. However, PR is not a complete solution: not all regions of the UK offer PR, PR only has on average a 50% uptake rate by patients and the drop-out rate is 30%. Also a significant proportion of patients (about 30%) do not increase their exercise capacity as a result of PR19, perhaps because breathlessness limits the training they complete or their peripheral muscle strength is normal19. Therefore, there is interest in alternative treatments or add-ons to exercise, particularly in terms of localised muscle treatments that are not limited by impaired respiratory function. Repetitive electrical stimulation of the femoral nerve (rES) appears to be an effective alternative method of passively training the quadriceps muscle. 30 minutes rES at 10Hz five times a week to both legs increased muscle strength and exercise performance in patients with COPD21 and those with heart failure22. Similar results have been achieved with fifteen minutes of repetitive magnetic stimulation of the femoral nerve (rMS) three times a week23. However, treatment studies with rES to investigate effects on exercise performance have often used separate treatment and control groups which introduces inter-subject differences into studies already limited by sample size243 and have only used voluntary measures of quadriceps function96. The only biopsy study of rES used a cross-over design but biopsies were only taken before and after the rES training period and not before and after the control period.244 The rMS study involved a total of eighteen subjects (ten assigned to rMS, eight to control) and biopsies were not taken to evaluate histological changes in the muscle. With this study, I sought primarily to evaluate the changes in quadriceps fibre characteristics as a result of an intensive rMS protocol, and secondarily, compare changes in quadriceps function as the result of rMS with the clinical gold standard for improving muscle function, PR.

Methods

Ethical approval The Research Ethics Committee of the Ealing & West London Mental Health Trust approved the study (06/Q0410/54). The trial was registered with National Clinical Trials Database (NCT 00737698). 2.13.1

Sample size calculation The sample size required for the training study was based on power calculations from a previous study on PR from our group221 and pilot data from our group on the effect of rMS on muscle strength (Swallow et al, unpublished) using Stata 10 statistical software. The power calculations were based on functional improvements (increase of 54m on 6MW as a result of PR and 10% increase in quadriceps TwQ as a result of rMS, as the minimum clinically significant increments) rather than increases in muscle fibre CSA or type I fibre proportions as the data for the latter was not available. We chose an increase of 10% twitch force as the minimally significant increment as previous data from Mador et al showed a 9.7% increase in twitch force as the result of 8 weeks PR17. A conventional power of 80% with a two-tailed p value of ≤0.05 was chosen indicating that a minimum of ten patients were required for the PR arm and twenty six for the rMS arm. We aimed to recruit fifteen to the PR group and thirty to the rMS group to allow for patient drop-out at the rates we have previously encountered. At completion, there were seventeen in the PR group and thirty seven in the rMS group.

Subject selection Eighty six COPD patients consented for the cross-sectional study also consented for the training study therefore the inclusion and exclusion criteria were as for the cross-sectional study. Patients were precluded from starting any new exercise regimen or new regular medication from consent to completion of the study, and patients were encouraged to contact me on day 1 of an acute exacerbation so appropriate treatment could be instituted. The study design and flow of participants through the study are shown in Fig. 4.1 and 4.2.

Randomisation FFMI was calculated using bioelectrical impedance (Methods chapter Section 2.4.2.1) and patients stratified into low FFMI (<15 kg/m2 for females, <16 kg/m2 for males) and normal FFMI. The low and normal FFMI groups were randomised separately (so low FFMI patients were evenly distributed between treatment groups) using a sealed envelope system and a block of 4 procedure weighted 2:1:1 for rMS: PR: no active treatment as the power calculation suggested that at least twice as many patients were required in the PR arm as the rMS arm.

Pre-training assessments Lung function, FFMI, quadriceps strength, quadriceps endurance, physical activity and 6MW and maximal cycle ergometry performance and HRQOL measurements were performed as described in the Methods chapter Sections 2.4-2.7. Percutaneous biopsy of the quadriceps and muscle fibre type analysis were performed. Patients underwent the pre-training physiological assessment and biopsies within four weeks of randomisation. The assessment was as described for the cross-sectional study (in the rMS group both legs were tested on the same day, in the other two groups the leg ipsilateral to the dominant hand was tested) and then patients proceeded to their allocated treatment within two weeks.

Training protocols

Repetitive magnetic stimulation of the femoral nerve (rMS) This was delivered using the Magstim Rapid magnetic nerve stimulator system (Magstim, Whitland Dyfed, UK) and supervised by myself at RBH Muscle Lab. The patient sat upright or reclined slightly backwards with the mat coil wrapped round the body of the quadriceps muscle to be trained, with the foot of the leg being stimulated positioned in a strap so that the contractions were isometric (Fig. 2.8). The stimulation frequency was 40Hz with a duty cycle of 0.4 (1s on, 4s off). Patients had three hours continuous rMS (apart from toilet breaks) twice a week over an 8-week period with at least twenty four hours rest between sessions. At the first session the stimulus intensity was increased from 22% power to 40% power, and subsequent sessions were at 40% power as this was the upper limit of what patients could tolerate and the machine could deliver for the whole session. 40% power generally generated between 10-20% of the patient's MVC.

Pulmonary Rehabilitation (PR) This was run by a research respiratory physiotherapist at the Royal Brompton Hospital twice a week with a maximum of three patients per session so training was closely supervised. Training consisted of a warm-up, then one hour aerobic work with subjects exercising on a stationery bicycle at a workload that produced 80% of their peak VO2 on a maximal incremental cycle ergometry protocol, on a treadmill, climbing stairs, and a combination of leg resistance exercises involving leg weights, squats and sit-to-stand manoeuvres, followed by a cool-down. Attempts were made at each session to increase the intensity and/or number of repetitions of each exercise. The exercise sheet used by the supervising physiotherapist to chart achievements is shown in Fig. 2.9.

No active treatment (Controls) Controls were asked to continue with their usual activities and were contacted by telephone two to three times during the 8-week period to minimise drop-out and to monitor for acute exacerbations of COPD. After study completion, these patients were enrolled on the PR course at RBH if they wished.

Post-training assessments For the PR and rMS groups, the physiological tests were done four to five days after the last training session, and three to four days later the biopsies were taken. Controls were assessed in the same week as the others. The timing was aimed at minimising group differences from varying delays between the last training session and testing. Post-training assessments involved all the same tests as the pre-training assessment.

Statistical analysis The primary outcomes measures were a) change in quadriceps fibre proportions and fibre CSA in trained leg versus untrained leg in rMS group and b) change in quadriceps function in rMS group versus PR group. All statistical analysis was performed using SPSS (SPSS 15, Chicago, USA). The Mann-Whitney U test was used to assess group differences (patients vs controls, trained vs untrained leg, change in trained leg vs change in untrained leg), Spearman's rank correlation coefficient was calculated to assess correlations and the Wilcoxon Signed-Ranks test used to examine differences between pre and post-training results in both the trained and the untrained leg (data not normally distributed). An interaction factor was calculated to assess the effect of exacerbation during the study. A two-tailed p value of ≤0.05 was used to define statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Cardiac failure
* Renal failure
* Liver failure
* Diabetes mellitus
* Systemic inflammatory diseases eg Rheumatoid arthritis, SLE
* Warfarin, coagulation problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Polkey, MBBSFRCPPhD, Study Director — Royal Brompton Hospital/Imperial College; Samantha A Sathyapala, MABMBChPhD, Principal Investigator — Imperial College London
Locations (1):
- Respiratory Muscle Lab, Royal Brompton Hospital, Fulham Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 86 enrolled and 71 completed the study
Groups:
- Repetitive Magnetic Stimulation: Repetitive magnetic stimulation
  Repetitive magnetic stimulation: Repetitive magnetic stimulation of the intramuscular branches of the femoral nerve for 3 hours twice a week for 8 weeks
Period: Overall Study
Arm/Group | Exercise | Repetitive Magnetic Stimulation | Control
Started | 23 | 42 | 21
Completed | 17 | 37 | 17
Not Completed | 6 | 5 | 4
Not completed — Withdrawal by Subject | 6 | 5 | 3
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Repetitive Magnetic Stimulation | Control | Total
Number analyzed (Participants) | 17 | 37 | 17 | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [63 to 77] | 66 [59 to 74] | 67 [61 to 74] | 67 [61 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 5 | 24
  Male | 10 | 25 | 12 | 47
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 37 | 17 | 71

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Fibre Size of Type IIa Fibres
Description: Quadriceps fibre cross-sectional area type II a fibres in quadriceps fibre.
Time Frame: 8 weeks
Population: Per protocol analysis
Measure: Median (Inter-Quartile Range); unit: micrometers squared
Arm/Group | Exercise | Repetitive Magnetic Stimulation | Control
Number analyzed (Participants) | 17 | 37 | 17
micrometers squared | 3885 [3175 to 4985] | 4326 [3299 to 5237] | 3610 [3168 to 4487]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Definition of adverse event and/or serious adverse event does not differ from clinicaltrials.gov definitions
Arm/Group | Exercise | Repetitive Magnetic Stimulation | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/42 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/42 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/42 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes